CLINICAL TRIAL: NCT05461378
Title: Prospective Observational Cohort Study of Pre-Exposure Prophylaxis of COVID-19 in Immunocompromised Patients Receiving the Monoclonal Antibody AZD7442 (EVUSHELD)
Brief Title: PREP (Pre-Exposure Prophylaxis) of COVID-19
Acronym: PrEP
Status: Completed | Type: Observational
Sponsor: Ghady Haidar (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Ghady Haidar, Assistant Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: PrEP C-19
Record Dates: First submitted 2022-07-12; First posted 2022-07-18 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Immuno-Deficiency; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — cilgavimab and tixagevimab drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, serum, and cellular components may be collected from whole blood samples. SARS-CoV-2 may be isolated from nasal and respiratory samples of persons with COVID-19. Investigators may also collect remnant swabs and blood from persons with COVID-19.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Outpatients: Outpatients who have not yet received EVUSHELD but who plan on receiving it in the future.
  Interventions: Drug: Evusheld
- Select inpatients (SOT/HCT/CAR-T): Newly transplanted adult solid organ transplant and HCT recipients, as well as CAR-T-cell therapy recipients, during their hospitalization to undergo SOT/HCT/CAR-T-cell therapy
  Interventions: Drug: Evusheld
- Individuals who have received EVUSHELD: Individuals who have received EVUSHELD within 9 months of enrollment.
  Interventions: Drug: Evusheld

INTERVENTIONS:
Drug: Evusheld — Participants who have received or plan to receive Evusheld.

SUMMARY:
This is a study of immunocompromised individuals who have received or plan to receive a drug called EVUSHELD. This study is looking at any serious adverse events that might happen after receiving EVUSHELD, the levels of EVUSHELD in participant's blood, blood antibody levels, neutralizing antibodies against SARS-CoV-2 (the virus that causes COVID-19), and other blood responses related to the immune system and COVID-19. Investigators are collecting blood and may also collect other samples such as nose swabs, oral swabs, or saliva.

DETAILED DESCRIPTION:
This is a prospective study of 500 immunocompromised participants at UPMC health system. EVUSHELD will be given according to the EUA in the United States as a part of standard of care by the patient's health care provider. Patients who receive intramuscular EVUSHELD as standard of care will be enrolled and followed for 12-months. The target sample size is 500 immunocompromised individuals; serum concentrations of AZD7442 will be obtained in all patients at the 6 (or at enrollment if the time point has passed) and 12 month timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 and at least 40 kg
* Eligible for EVUSHELD as per the EUA

Exclusion Criteria:

* Active and confirmed COVID-19
* Known or suspected pregnancy, concurrent lactation
* Any other significant disease, disorder, or finding, in the opinion of the investigator, that may significantly increase the risk to the participant because of participation in the study, affect the ability of the subject to participate in the study, or impair interpretation of the study data

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Immunocompromised Patients using the Monoclonal Antibody EVUSHELD (AZD7442)
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Concentration of AZD7442 in serum over time [ENROLLMENT, 6 MONTHS, 12 MONTHS] Concentration of AZD7442 in serum over time [ENROLLMENT, 6 MONTHS, 12 MONTHS] Concentration of AZD7442 in serum over time [ENROLLMENT, 6 MONTHS, 12 MONTHS] | 12-months
  The primary objective of PrEP C-19 is to measure AZD7442 serum concentration levels by blood draws at 6 months (or at enrollment if the time point has passed) and 12 months after IM administration of EVUSHELD.

SECONDARY OUTCOMES:
Concentration of AZD7442 in serum | 12-months
  Collected at 1, 3, AND 9 months
Assessment of SARS-CoV-2 Spike IgG levels using Bioplex/Biorad assays, viral neutralization assay using competitive ACE2 EIA, and pseudovirus neutralization titers | 12-months
  Collected at enrollment and 1, 3, 6, 9, and 12 months
Assessment of T-cell responses using an ELISPOT assay | 12-months
  Obtained before and after vaccination
Determining SARS_CoV-2 variant type using whole genome sequencing | 12-months
  Collected among subjects with breakthrough infection
Determining Concentration of AZD7442 in serum, SARS-CoV-2 Spike IgG levels using Bioplex/Biorad assays, viral neutralization assay using competitive ACE2 EIA, and pseudovirus neutralization titers | 12-months
  Collected during breakthrough infection
Proportion of participants with ≥1 COVID-19-related medically-attended visit | 12-months
  Participants with ≥1 COVID-19-related medically-attended visit
Proportion of participants who die by the end of the study | 12-months
  COVID-19 associated and all-cause mortality
Lifestyle Modification Questionnaire | 12-months
  Proportion of participants who report changes in lifestyle

CONTACTS AND LOCATIONS:
Overall Officials: Ghady Haidar, MD, Principal Investigator — University of Pittsburgh and UPMC
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Share study reports to AstraZeneca, de-identified data only will be shared